CLINICAL TRIAL: NCT02975583
Title: A Double-blind, Randomized, Parallel Design Two Center Study to Compare the Effect of Vorapaxar vs. Placebo on Lower Extremity Vein Graft Maturation, Remodeling, and Function
Brief Title: Vorapaxar and Lower Extremity Bypass Grafts
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We could not secure adequate medication
Sponsor: Vanderbilt University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joshua Beckman, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 161925
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Artery Disease
Keywords: Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis | interventions — vorapaxar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Vorapaxar (Active Comparator): Drug: Vorapaxar 2.08 mg orally daily for a year Other name: Zontivity
  Interventions: Drug: Vorapaxar
- Placebo Comparator: Placebos (Placebo Comparator): Medication: Matching Placebo Daily tablet
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Vorapaxar — 2.08 mg oral tablet daily
  Other Names: Zontivity
  Arms: Experimental: Vorapaxar
Drug: Placebos — Placebo oral tablet daily
  Other Names: Placebo
  Arms: Placebo Comparator: Placebos

SUMMARY:
There are no medical therapies indicated for reduction of limb ischemic events. Studies of dual-antiplatelet therapy with aspirin and clopidogrel versus aspirin alone (CASPAR) as well as studies of systemic anticoagulation (WAVE) have shown no benefit for either strategy in the reduction in limb vascular events. Surgical bypass grafting involves harvesting of the vein, warm ischemia with disruption of vaso vasorum, ischemia-reperfusion, and finally heightened hemodynamic stress in the new arterial environment. Vein grafts rapidly remodel in response to the increase in blood flow and pressure in an attempt to normalize them into physiological range. The investigators have previously identified 3 distinct temporal phases of the remodeling process: During the first 30 days following implantation is a critical period of luminal enlargement which appears to be an endothelium-independent process. The second phase occurs between 1 and 3 months and represents a period of stiffening of the vein graft indicating synthesis of fibrous proteins. The third period is referred to as biochemical remodeling wherein the vein recovers clinically measureable endothelial function. It is likely diabetes mellitus impacts each of these phases. TRA2°P-TIMI 50 demonstrated a reduction in acute limb ischemic (ALI) events (42% reduction) and urgent peripheral arterial revascularizations (35% reduction), a finding unique among medical therapies. While the temporal trend in reduction in ALI events occurred early and late after exposure suggestion an antithrombotic mechanism, the reduction in elective revascularization occurred later suggested beneficial effects beyond platelet inhibition. The purpose of this trial is to study the physiological impact of vorapaxar on lower extremity bypass graft maturation and function.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is characterized by atherosclerotic occlusive disease of the lower extremities. More than 8 million Americans and 200 million people globally have PAD. Recent data reveal a prevalence of 15% in the MEDICARE population. In populations at risk, patients with a history of diabetes or cigarette smoking, the risk may rise as high as 30%. In addition to the heightened risk of myocardial infarction and stroke, PAD increases the risk of lower extremity claudication and critical limb ischemia. Lower extremity bypass grafting is an important method of restoring blood flow to the distal limb, reducing symptoms of claudication, and preventing amputation in patients with severe PAD.

Vorapaxar is a protease activated receptor (PAR)-1 antagonist that inhibits thrombin activation of the PAR-1 receptor. Vorapaxar has been FDA approved for patients with PAD to reduce the rate of cardiovascular death, MI, stroke, and urgent coronary revascularization. It is prohibited in patients with a previous stroke. In addition, patients treated with vorapaxar were noted to have a significant reduction in the rates of acute limb ischemia. This study will be a randomized, double blind, placebo-controlled randomized study of vorapaxar vs. placebo in 80 patients undergoing femoral-popliteal bypass grafting for Rutherford 3 - 5 disease.

Baseline visit: Informed consent will be signed. Vital signs will be taken and blood drawn fasting for baseline values.

First visit, pre-surgery: Blood will be drawn for platelet activation testing. A 6 minute walk test will be performed. Brachial artery reactivity testing will be performed. An ankle-brachial index will be performed.

30 days: Platelet testing will be performed. 90 days: Limited history and physical exam. 180 days: Limited history and exam, blood draw for biomarkers, brachial artery reactivity testing. Vein bypass graft reactivity testing.

360 days: 6 minute walk test and ankle brachial index will be performed.

Randomization: The Investigational Pharmacy will create a block randomization. Patients in the active treatment group will receive vorapaxar 2.08 mg daily or matching placebo. Treatment will continue for 1 year.

In addition, 20 healthy subjects to serve as a control population to define normal parameters during a single visit day. The healthy subjects will not be administered vorapaxar or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 35 years or older
* Atherosclerotic, infrainguinal PAD
* Rutherford classes 3-5 planned for lower extremity bypass grafting
* Adequate inflow into the index femoral artery
* Adequate popliteal, tibial, or pedal revascularization target
* Willing to comply with protocol, attend follow-up appointments, complete all study assessments, and provide informed consent

Exclusion Criteria:

* Complete occlusion of the iliac artery
* Aortoiliac occlusive disease or severe common femoral artery disease
* Presence of a femoral, popliteal or tibial aneurysm of the index limb
* Life expectancy less than 2 years
* A vascular disease prognosis that includes an anticipated above ankle amputation on index limb within 4 weeks of index procedure
* Renal dysfunction defined as MDRD eGFR ≤ 30ml/min/173 m2 at the time of screening
* Currently on dialysis or history of a renal transplant
* A documented hypercoagulable state
* Nonatherosclerotic occlusive disease
* Any prior infrainguinal revascularization
* Current immunosuppressive medication, chemotherapy or radiation therapy
* Absolute contraindication to iodinated contrast
* Women who are pregnant
* Women who are nursing

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Bypass Graft Flow Mediated Vasodilation under Fasted Conditions using B-mode ultrasonography on Day 180 for each treatment condition. | 6 Months
  Ultrasonographic evaluation of the graft before and after sphygmomanometric cuff inflation on the calf is performed and the measure of interest is percent increase in vein graft diameter.

SECONDARY OUTCOMES:
Change From Baseline in Flow Mediated Vasodilation (FMD) Under Fasted Condition on Day 180 [ Time Frame: baseline and day 180 for each treatment arm ] | 6 Months
  Ultrasonographic evaluation of the graft before and after sphygmomanometric cuff inflation on the arm is performed and the measure of interest is percent increase in brachial artery diameter.
Platelet Activation blood testing | 30 days
  The investigators will be measuring levels of platelet dilysyl-MDA cross-links 30 days after treatment initiation. Higher levels indicate more platelet activation.
Change in Six Minute Walk Test from Baseline to 1 year | One year
  The distance walked in a 100 foot hallway in 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Beckman, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.